CLINICAL TRIAL: NCT03779204
Title: Transitioning Youth Out of Homelessness: A Mixed Methods Community-Based Pilot Randomized Controlled Trial of a Rent Subsidy and Mentoring Intervention in Three Canadian Cities
Brief Title: Effect of a Rent Subsidy and Mentoring on Youth Transitioning Out of Homelessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Covenant House Toronto (Other); Living Rock Ministries (Other); Resource Association for Teens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-251
Record Dates: First submitted 2018-09-23; First posted 2018-12-19 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-09

CONDITIONS: Homeless Persons
Keywords: Social Isolation; Self-Esteem; Hope; Psychiatric Problem; Education; Employment; Income; Housing Problems; Identity, Social; Youth; Rent Subsidy; Mentorship
MeSH Terms: conditions — Social Isolation; Social Identification

STUDY DESIGN:
Intervention Model Description: This study will employ a convergent mixed methods design (i.e., quantitative and qualitative data are collected concurrently, and the findings combined) embedded within a RCT and a CBPAR framework. 24 participants will be assessed for eligibility, and then randomized into 1 of 2 arms using covariate adaptive randomization. 12 are allocated to the intervention group (rent subsidies + mentoring), while 12 are allocated to the control group (rent subsidies only). Participants in the intervention group (n = 12) will be matched with an adult mentor recruited by one of the community partners. Mentors are selected and matched through one-on-one interviews with someone in a leadership role within the organization. A common mentoring guide will be used for all sites; these booklets cover information ranging from ideal mentor characteristics to mentor code of conduct.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rent subsidies + Mentorship (Experimental): Participants in this arm (n = 13) will receive rent subsidies (ranging from $400 - $500/month) for 24 months as part of the intervention and be matched with an adult mentor recruited by one of the community partners.
  Interventions: Behavioral: Mentorship; Behavioral: Rent Subsidies
- Rent subsidies only (Active Comparator): Participants in this arm (n = 11) will receive rent subsidies only (ranging from $400 - $500/month) for 24 months as part of the comparator group intervention. This group will not receive mentorship.
  Interventions: Behavioral: Rent Subsidies

INTERVENTIONS:
Behavioral: Mentorship — The mentors will be encouraged to incorporate the key relationship-based components of natural mentors (e.g., a 'coach' or 'cheerleader' role) to assist with mainstream integration. The mentors will have more flexibility than a typical formal mentorship program in the types of activities they pursue with their mentees. They will not be mandated to attend shelter-based social events, but rather engage in activities that direct their mentees away from the shelter system (and their old identities as homeless youth) and toward the mainstream (e.g., meeting for coffee at a local university campus). All of the mentors will meet monthly with their mentees for two years. In addition, the mentor will be encouraged to touch base with their mentee via phone or text message every week. If a mentor is unable to continue their role and there are at least six months left in the study, the study participant will be matched with a new mentor.
  Arms: Rent subsidies + Mentorship
Behavioral: Rent Subsidies — Participants will receive rent subsidies ($500 for those living in Toronto, $400 for those living in Hamilton or St. Catherine's due to differences in cost of living) for 24 months.

SUMMARY:
Compared to the vast amount of literature about the risk factors associated with young people entering and becoming entrenched in homelessness, much less is known about how to facilitate and sustain transitions off the streets.

Current evidence indicates that while structural supports such as subsidized housing and social service providers are important, these things alone are insufficient to help young people integrate into mainstream society. Connecting these young people with an adult who exhibits the relationship-based components of mentoring that young people value most (e.g., genuine interest in their well-being and belief in their ability to succeed, a non-judgmental attitude and a willingness to listen, the provision of advice, guidance, affirmation and encouragement) may be key to helping them move forward and integrate into the mainstream.

This intervention will provide 24 young people (ages 18-26) who have transitioned out of homelessness and into market rent housing within the past year with rent subsidies for 24 months. Half of the young people will be randomized to receive regular mentorship from an adult mentor, tasked with helping their mentee bridge the gap between homelessness and mainstream living.

It is hypothesized that, for the primary outcome measures of community integration and self-esteem:

1. Better mean scores (community integration and self-esteem) in the participants who receive rent subsidies plus mentorship (intervention group) will be observed compared to the participants who receive rent subsidies only (control group) by the primary endpoint of 18 months of study participation.

It is hypothesized that, for the secondary outcome measures of social connectedness, hope, and academic and vocational participation:

1. Better mean scores (social connectedness and hope) in the intervention group relative to participants in the control group will be observed by 18 months of study participation.
2. Participants in the intervention group will be more likely than the control group to demonstrate sustained engagement in academic and vocational activities (education, employment, and/or skills training) by 18 months of study participation.

This pilot will be the first to test the impact of economic and social supports on meaningful social integration for formerly homeless young people living in market rent housing.

DETAILED DESCRIPTION:
The overarching aim of this mixed methods study is to assess whether and how rent subsidies and mentorship influence social integration outcomes for formerly homeless young people living in market rent housing in three urban settings.

Specifically, the objectives of this study are to:

1. Determine whether rent subsidies plus mentorship results in better social integration outcomes than only receiving rent subsidies with respect to: a) community integration (psychological and physical); and b) self-esteem at the primary endpoint of 18 months.
2. Determine whether rent subsidies plus mentorship results in better social integration outcomes than only receiving rent subsidies with respect to: a) social connectedness; b) hope; and c) sustained academic and vocational participation at 18 months.
3. Explore whether rent subsidies plus mentorship results in better social integration outcomes than only receiving rent subsidies with respect to: a) income; b) perceived housing quality; c) psychiatric symptoms; and d) sense of engulfment at 18 months.
4. Integrate qualitative data to facilitate a fuller understanding of the quantitative data and deepen understanding of what the study participants (young people and mentors) found most beneficial about the intervention and how it could be improved.

This study will employ a convergent mixed methods design (i.e., quantitative and qualitative data are collected concurrently, and the findings combined) embedded within a randomized controlled trial (RCT) and a community-based participatory action research (CBPAR) framework. A mixed methods RCT is appropriate given the complex explanatory pathways (i.e., social and behavioral processes that may act independently and interdependently) of this intervention. In addition, the qualitative data will provide insights on contextual factors that may impact the external validity of the findings. Most importantly, this design provides a crucial (and under utilized) youth-informed perspective on social integration.

The study will be conducted in three Canadian cities: Toronto, Ontario (pop. 2.8 million); Hamilton, Ontario (pop. 552,000); and St. Catharines, Ontario (pop. 133,000). All of the study participants (n = 24) will receive rent subsidies (ranging from $400 - $500/month) for 24 months as a part of the intervention. This study includes funding for the rent subsidies and will be paid directly to the landlords by the community partners. St. Michael's Hospital will establish a service provider agreement with each of the community partners for this purpose. Participants in the intervention group (n = 12) will be matched with an adult mentor recruited by one of the community partners.

The mentors will be encouraged to incorporate the key relationship-based components of natural mentors (e.g., a 'coach' or 'cheerleader' role) to assist with mainstream integration. To facilitate more of an organic, natural mentor-mentee relationship, the mentors will have more flexibility than a typical formal mentorship program in the types of activities they pursue with their mentees. For example, they will not be mandated to attend shelter-based social events. Instead, mentors will be encouraged to initiate activities that direct their mentees away from the shelter system (and their old identities as homeless youth) and toward the mainstream (e.g., meeting for coffee at a local university campus, touring a local library, or visiting the mentor's place of employment during business hours). All of the mentors will meet monthly with their mentees for two years. In addition, the mentor will be encouraged to touch base with their mentee via phone or text message every week. If a mentor is unable to continue their role and there are at least six months left in the study, the study participant will be matched with a new mentor.

Community partners will match all participants with an outreach worker (already employed by each agency) who will communicate regularly with the research team, help ensure the rent subsidies are being distributed appropriately, maintain an ongoing relationship with the study participants, and monitor for 'red flags' in participants matched in mentor-mentee relationships (e.g., mentee reluctant to meet with their mentor). Matching all of the study participants with a worker will also help ensure that everyone is receiving a fairly equal level of social support from community partners, making it easier for the research team to discern whether the outcomes of interest are more likely attributable to mentorship rather than to varied levels of agency-based support. Moreover, a review of services and interventions designed to reduce "problem behaviors" (e.g., substance use and risky sexual practices) among street-involved and homeless young people (ages 12 - 24) found that researchers who had strong relationships with outreach workers and the community had more effective interventions and lower attrition rates than those who did not.

Following the baseline interview, participants at each of the three study sites (Toronto (n=12), Hamilton (n=6), and St. Catharine's (n=6)) will be randomized using block randomization to either the intervention (rent subsidies plus mentoring) or control (rent subsidies only) group. Randomization will be balanced by site based on random block sizes of two and four. The advantage of using block randomization is to uniformly distribute participants into treatment groups within each site. Because small block sizes may increase the risk of guessing the allocation procedure and subsequently introducing bias into the enrolment procedure, random block sizes will be used to avoid this potential selection bias. A unique randomization schedule will be produced for each site using SAS. A research coordinator not affiliated with the study will be the only person with access to the randomization schedule. The research coordinator will prepare sealed, opaque and sequentially numbered envelopes with the randomization results of participants. After assessing for eligibility and obtaining consent of each participant, research personnel responsible for enrolling participants will open the next randomization envelope from the sequentially ordered randomization envelope file to obtain the participant's randomized group assignment.

Quantitative data will be collected at six points in time over the course of 30 months: baseline, month six, month 12, month 18, month 24, and month 30. Qualitative measures are an important feature of this study and will consist of: 1) semi-structured individual interviews (study participants) and 2) focus groups (mentors). At baseline, twelve participants (six from each arm of the study) will be invited to participate in six semi-structured individual interviews, which will take place at the same time as the quantitative data collection: baseline, month six, month 12, month 18, month 24, and month 30. Participants will be purposively selected with a goal of having input from each of the three communities and a fairly equal gender and ethno-racial representation. All of the mentors (n = 12) will be invited to participate in two focus groups, which will take place at month 12 and month 24.

All analyses will be performed using the intention-to-treat principle; that is, all participants will be included and analyzed in the groups they were originally randomized. Baseline characteristics of the intervention and control groups will be summarized using descriptive statistics (i.e., mean, standard deviation, median and interquartile range for continuous variables, and frequencies and proportions for categorical variables). The descriptive statistics for outcomes at each study time point will be calculated, and differences in trajectories from baseline to 30 months follow-up between intervention and control groups using scatterplots and box-plots will be explored. Differences with 95% confidence intervals in continuous outcomes at 18 months (psychological community integration, self-esteem, social connectedness, hope, perceived housing quality, psychiatric symptoms, and sense of engulfment) between participants who received rent subsidies plus mentorship and participants who only received rent subsidies will be estimated using Analysis of Covariance (i.e., linear regression models), including an indicator of intervention group and the baseline value of the outcome. Regression diagnostics will be performed and analyses using the non-parametric Wilcoxon rank-sum test will be repeated if there are extreme outliers or influential observations. Groups will be compared with respect to count outcomes at 18 months (physical community integration) using graphical tools and the non-parametric Wilcoxon rank-sum test. For binary outcomes at 18 months (sustained academic and vocational participation, and income above low income cut-off ), differences in proportions with 95% confidence intervals will be estimated and tested using the chi-square or Fisher's exact test. Given the small sample size of this pilot randomized trial, all results will be interpreted with caution and with the intention of generating data and hypotheses for conducting a larger trial.

Given the emergent, iterative nature of research using a qualitative design, data analysis and interpretation will begin immediately after the first qualitative data generation session (at baseline). The semi-structured individual interviews and focus groups will be audio recorded and transcribed verbatim. In order to conduct a more nuanced analysis of the data, the transcriptionist will be instructed to note short responses, uncooperative tones, and literal silence. Prior to each subsequent qualitative data generation session, members of the research team will conduct a preliminary data analysis, reading the interview transcripts multiple times, separating the data into coded segments, making analytic memos beside sections of the transcripts, identifying emerging themes (and comparing/contrasting these between respondents), and compiling new questions. Those participating in the individual interviews and the focus groups will be asked for their perspectives on the emerging interpretations at each visit and these perspectives will play a key role in helping shape the data analysis and help ensure the trustworthiness of the data. The web-based application Dedoose will be utilized to assist with sorting and coding the qualitative data.

In keeping with CBPAR methodology, disseminating evidence with community partners is key in building community capacity and improving the lives of the young people participating in this study. Moreover, given the use of Critical Social Theory, the study findings will not only be presented, but will also be used to expose and explicate the relational processes (e.g., subjective experience of low socioeconomic position and low social class) that may be preventing formerly homeless young people from achieving meaningful social integration. With an emphasis on 'actionable' data, the findings will be disseminated broadly to both academic and community-based audiences in a variety of formats ranging from scientific journal papers to oral presentations.

ELIGIBILITY:
Inclusion Criteria:

* Be between ages 18-26
* Left homelessness within the past year
* Living in market rent housing
* Plan on staying in or nearby the community in which they were recruited (Toronto, Hamilton, or St. Catharines) for the duration of the 24-month study
* Be willing to be matched with an adult mentor who has been screened and chosen by one of the community partners

Exclusion Criteria:

* In imminent danger of losing their housing (e.g., facing jail time or impending eviction)
* Enrolled in another study with enhanced financial and social supports
* Unable to provide free and informed consent
* Unable to communicate fluently in English

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi S Thulien, RN, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Altena AM, Brilleslijper-Kater SN, Wolf JL. Effective interventions for homeless youth: a systematic review. Am J Prev Med. 2010 Jun;38(6):637-45. doi: 10.1016/j.amepre.2010.02.017. PMID 20494240
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Background] Brueckner, M., Green, M., & Saggers, S. (2011). The trappings of home: Young homeless people's transitions towards independent living. Housing Studies, 26(1), 1-16. doi:10.1080/02673037.2010.512751.
- [Background] Chenail. R. J., St. Goerge, S., Wulff, D., & Cooper, R. (2012). Action research: The methodologies. In P. L. Munhall (Ed.), Nursing research: A qualitative perspective (5th ed.) (pp. 455-470). Sudbury, MS: Jones & Bartlett.
- [Background] Ciarolo, J. A., Edwards, D. W., Kiresuk, T. J., Newman, F. L., & Brown, T. R. (1981). Colorado symptom index. Washington, DC: National Institute of Mental Health.
- [Background] Coren E, Hossain R, Pardo Pardo J, Bakker B. Interventions for promoting reintegration and reducing harmful behaviour and lifestyles in street-connected children and young people. Cochrane Database Syst Rev. 2016 Jan 13;2016(1):CD009823. doi: 10.1002/14651858.CD009823.pub3. PMID 26760047
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Creswell, J.W. (2014). Research design: Qualitative, quantitative, and mixed method approaches (4th ed.). Thousand Oaks, CA: Sage.
- [Background] Creswell, J.W., & Plano Clark, V.L. (2018). Designing and conducting mixed methods research (3rd ed.). Thousand Oaks, CA: Sage.
- [Background] Dang MT, Miller E. Characteristics of natural mentoring relationships from the perspectives of homeless youth. J Child Adolesc Psychiatr Nurs. 2013 Nov;26(4):246-53. doi: 10.1111/jcap.12038. Epub 2013 Jun 14. PMID 24180604
- [Background] Denzin, N.K., & Lincoln, Y.S. (2011). The SAGE handbook of qualitative research. Thousand Oaks, CA: SAGE Publications Inc.
- [Background] Eakin JM, Mykhalovskiy E. Reframing the evaluation of qualitative health research: reflections on a review of appraisal guidelines in the health sciences. J Eval Clin Pract. 2003 May;9(2):187-94. doi: 10.1046/j.1365-2753.2003.00392.x. PMID 12787182
- [Background] Farquhar MC, Ewing G, Booth S. Using mixed methods to develop and evaluate complex interventions in palliative care research. Palliat Med. 2011 Dec;25(8):748-57. doi: 10.1177/0269216311417919. Epub 2011 Aug 1. PMID 21807749
- [Background] Fletcher, R.H., Fletcher, S.W., & Fletcher, G.S. (2014). Clinical epidemiology: The essentials (5th ed.). Philadelphia, PA: Lippincott Williams & Wilkins.
- [Background] Frederick, T., Chwalek, M., Hughes, J., Karabanow, J., & Kidd, S. (2014). How stable is stable? Defining and measuring housing stability. Journal of Community Psychology, 42(8), 964- 979. doi:10.1002/jcop.21665.
- [Background] Gaetz, S. (2014). Coming of age: Reimagining the response to youth homelessness in Canada. Toronto, ON: The Canadian Homelessness Research Network Press. Retrieved from http://www.homelesshub.ca/comingofage
- [Background] Gaetz, S., Dej, E., Richter, T., & Redman, M. (2016) The state of homelessness in Canada 2016. Toronto, ON: Canadian Observatory on Homelessness Press. Retrieved from http://www.homelesshub.ca/SOHC2016
- [Background] Gaetz, S., O'Grady, B., Kidd, S., & Schwan, K. (2016). Without a home: The national youth homelessness survey. Toronto: Canadian Observatory on Homelessness Press. Retrieved from http://homelesshub.ca/sites/default/files/WithoutAHome-final.pdf
- [Background] Gaetz, S., & Redman, M. (2016). Federal investment in youth homelessness: Comparing Canada and the United States and a proposal for reinvestment. Canadian observatory on homelessness policy brief. Toronto, ON: The Homeless Hub Press. Retrieved from http://homelesshub.ca/sites/default/files/Policy_Brief.pdf
- [Background] Goodkind JR, Amer S, Christian C, Hess JM, Bybee D, Isakson BL, Baca B, Ndayisenga M, Greene RN, Shantzek C. Challenges and Innovations in a Community-Based Participatory Randomized Controlled Trial. Health Educ Behav. 2017 Feb;44(1):123-130. doi: 10.1177/1090198116639243. Epub 2016 Jul 10. PMID 27179291
- [Background] Hammersley, M., & Atkinson, P. (2007). Ethnography: Principles in Practice (3rd ed.). London, UK: Routledge.
- [Background] Hwang SW, Burns T. Health interventions for people who are homeless. Lancet. 2014 Oct 25;384(9953):1541-7. doi: 10.1016/S0140-6736(14)61133-8. PMID 25390579
- [Background] Israel, B.A., Schulz, A.J., Parker, E.A., Becker, A.B., Allen, III, Guzman, R.J., & Lichtenstein, R. (2018). Critical issues in developing and following CBPR principles. In N. Wallerstein, B. Duran, J. Oetzel, & M. Minkler (Eds.), Community-based participatory research for health: Advancing social and health equity (3rd ed.) (pp. 31-44). San Francisco, CA: Jossey-Bass
- [Background] Karabanow, J. (2008). Getting off the street: Exploring the process of young people's street exits. American Behavioral Scientist, 51(6), 772-788. doi:10.1177/0002764207311987.
- [Background] Karabanow, J., Carson, A., & Clement, P. (2010). Leaving the streets: Stories of Canadian youth. Halifax, NS: Fernwood Publishing.
- [Background] Karabanow, J., Kidd, S., Frederick, T., & Hughes, J. (2016). Toward housing stability: Exiting homelessness as an emerging adult. Journal of Sociology & Social Welfare, 43(1), 121- 148. Retrieved from https://wmich.edu/socialworkjournal
- [Background] Kawabata, M., & Gastaldo, D. (2015). The less said, the better: Interpreting silence in qualitative research. International Journal of Qualitative Research Methods, 14(4), 1-9. doi:10.1177/1609406915618123.
- [Background] Kidd, S.A., Frederick, T., Karabanow, J., Hughes, J., Naylor, T., & Barbic, S. (2016). A mixed methods study of recently homeless youth efforts to sustain housing and stability. Child and Adolescent Social Work Journal, 33(3), 207-218. doi:10.1007/s10560-015-0424.
- [Background] Kozloff N, Adair CE, Palma Lazgare LI, Poremski D, Cheung AH, Sandu R, Stergiopoulos V. "Housing First" for Homeless Youth With Mental Illness. Pediatrics. 2016 Oct;138(4):e20161514. doi: 10.1542/peds.2016-1514. PMID 27681009
- [Background] Kulik DM, Gaetz S, Crowe C, Ford-Jones EL. Homeless youth's overwhelming health burden: A review of the literature. Paediatr Child Health. 2011 Jun;16(6):e43-7. doi: 10.1093/pch/16.6.e43. PMID 22654549
- [Background] Kusenbach, M. (2003). Street phenomenology: The go-along as ethnographic research tool. Ethnography, 4(3), 455-485. doi: 10.1177/146613810343007.
- [Background] Lee, R. M., & Robbins S. B. (1995). Measuring belongingness: The social connectedness and the social assurance scales. Journal of Counseling Psychology, 42(2), 232-241. doi: 10.1037/0022-0167.42.2.232.
- [Background] Lewin S, Glenton C, Oxman AD. Use of qualitative methods alongside randomised controlled trials of complex healthcare interventions: methodological study. BMJ. 2009 Sep 10;339:b3496. doi: 10.1136/bmj.b3496. PMID 19744976
- [Background] Loiselle, C.G., Profetto-McGrath, J., Polit, D.F., & Tatano Beck, C.T. (2004). Canadian essentials of nursing research. Philadelphia, PA: Lippincott Williams & Wilkins.
- [Background] Luchenski S, Maguire N, Aldridge RW, Hayward A, Story A, Perri P, Withers J, Clint S, Fitzpatrick S, Hewett N. What works in inclusion health: overview of effective interventions for marginalised and excluded populations. Lancet. 2018 Jan 20;391(10117):266-280. doi: 10.1016/S0140-6736(17)31959-1. Epub 2017 Nov 12. PMID 29137868
- [Background] Madison, D.S. (2012). Critical ethnography: Method, ethics, and performance (2nd ed.). Thousand Oaks, CA: Sage Publication, Inc.
- [Background] Mayock, P., O'Sullivan, E., & Corr, M.L. (2011). Young people exiting homelessness: An exploration of process, meaning and definition. Housing Studies, 26(6), 803-826. doi:10.1080/02673037.2011.593131.
- [Background] McCay, E., Carter, C., Aiello, A., Quesnel, S., Langley, J., Hwang, S., .... Karabanow, J. (2015). Dialectical Behavior Therapy as a catalyst for change in street-involved youth: A mixed methods study. Children and Youth Services Review, 58, 187-199. doi: 10.1016/j.childyouth.2015.09.021.
- [Background] Milburn NG, Rice E, Rotheram-Borus MJ, Mallett S, Rosenthal D, Batterham P, May SJ, Witkin A, Duan N. Adolescents Exiting Homelessness Over Two Years: The Risk Amplification and Abatement Model. J Res Adolesc. 2009 Dec 1;19(4):762-785. doi: 10.1111/j.1532-7795.2009.00610.x. PMID 25067896
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Ontario Human Rights Commission. (n.d.). Housing as a human right. Retrieved from http://www.ohrc.on.ca/en/right-home-report-consultation-human-rights-and-rental-housing-ontario/housing-human-right
- [Background] Popay, J., Escorel, S., Hernandez, M., Johnston, H., Mathieson, J., & Rispel, L. (2008). Understanding and tackling social exclusion: Final report to the WHO commission on social determinants of health from the social exclusion knowledge network. Retrieved from http://www.who.int/social_determinants/themes/socialexclusion/en/
- [Background] Prasad, P. (2005). Crafting qualitative research: Working in the postpositivist traditions. New York, NY: M.E. Sharpe.
- [Background] Public Interest. (2009). Changing patterns for street involved youth. Toronto, ON: Author. Retrieved from http://www.worldvision.ca/Programs-and- Projects/Canadian Programs/Documents/ChangingPatternsForStreetInvolvedYouth.pdf
- [Background] Quilgars, D., & Pleace, N. (2016). Housing First and Social Integration: A Realistic Aim? Social Inclusion, 4(4), 5-15. doi:10.17645/si.v4i4.672.
- [Background] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton, NJ: Princeton University Press.
- [Background] Rutman, A., Hubberstey, A., Barlow, A., & Brown, E. (2005). Supporting young people's transitions from care: Reflections on doing participatory action research with youth from care. In L. Brown & S. Strega (Eds.), Research as resistance: Critical, Indigenous, & anti-oppressive approaches (pp. 153-179). Toronto, ON: Canadian Scholars' Press/Women's Press.
- [Background] Slesnick N, Dashora P, Letcher A, Erdem G, Serovich J. A Review of Services and Interventions for Runaway and Homeless Youth: Moving Forward. Child Youth Serv Rev. 2009 Jul;31(7):732-742. doi: 10.1016/j.childyouth.2009.01.006. PMID 20161294
- [Background] SocioCultural Research Consultants, LLC. (2018). Dedoose (Version 8.0.35) [web application]. Retrieved from http://www.dedoose.com
- [Background] Solar, O., & Irwin, A. (2010). A conceptual framework for action on the social determinants of health: Social determinants of health discussion paper 2. Geneva, Switzerland: World Health Organization Press. Retrieved from http://www.who.int/sdhconference/resources/ConceptualframeworkforactiononS DH_eng.pdf
- [Background] Solomon, P., Cavanaugh, M.M., & Draine, J. (2009). Randomized controlled trials: Design and implementation for community-based psychosocial interventions. New York, NY: Oxford University Press.
- [Background] Stergiopoulos V, Gozdzik A, O'Campo P, Holtby AR, Jeyaratnam J, Tsemberis S. Housing First: exploring participants' early support needs. BMC Health Serv Res. 2014 Apr 13;14:167. doi: 10.1186/1472-6963-14-167. PMID 24725374
- [Background] Strega, B. (2005). The view from the poststructural margins: Epistemology and methodology reconsidered. In L. Brown & S. Strega (Eds.), Research as resistance: Critical, Indigenous, & anti-oppressive approaches (pp. 199-235). Toronto, ON: Canadian Scholars' Press/Women's Press.
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Thompson, A. E., Greeson, J. K., & Brunsink, A. M. (2016). Natural mentoring among older youth in and aging out of foster care: A systematic review. Children and Youth Services Review, 61, 40-50. doi: 10.1016/j.childyouth.2015.12.006.
- [Background] Thulien NS, Gastaldo D, Hwang SW, McCay E. The elusive goal of social integration: A critical examination of the socio-economic and psychosocial consequences experienced by homeless young people who obtain housing. Can J Public Health. 2018 Feb;109(1):89-98. doi: 10.17269/s41997-018-0029-6. PMID 29981071
- [Background] Toro PA, Passero Rabideau JM, Bellavia CW, Daeschler CV, Wall DD, Thomas DM, Smith SJ. Evaluating an intervention for homeless persons: results of a field experiment. J Consult Clin Psychol. 1997 Jun;65(3):476-84. doi: 10.1037//0022-006x.65.3.476. PMID 9170771
- [Background] Urbaniak, G.C., & Plous,S. (2013). Research Randomizer (Version 4.0) [Computer software]. Retrieved from https://www.randomizer.org
- [Background] Van Dam L, Smit D, Wildschut B, Branje SJT, Rhodes JE, Assink M, Stams GJJM. Does Natural Mentoring Matter? A Multilevel Meta-analysis on the Association Between Natural Mentoring and Youth Outcomes. Am J Community Psychol. 2018 Sep;62(1-2):203-220. doi: 10.1002/ajcp.12248. Epub 2018 Apr 25. PMID 29691865
- [Background] Wallerstein NB, Duran B. Using community-based participatory research to address health disparities. Health Promot Pract. 2006 Jul;7(3):312-23. doi: 10.1177/1524839906289376. Epub 2006 Jun 7. PMID 16760238
- [Background] Wallerstein N, Duran B. Community-based participatory research contributions to intervention research: the intersection of science and practice to improve health equity. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S40-6. doi: 10.2105/AJPH.2009.184036. Epub 2010 Feb 10. PMID 20147663
- [Background] Wallerstein, N., Duran, B., Oetzel, J.G., & Minkler, M. (2018). Community-based participatory research for health: Advancing social and health equity (3rd ed.). San Francisco, CA: Jossey-Bass.
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Result] Thulien NS, Amiri A, Hwang SW, Kozloff N, Wang A, Akdikmen A, Roglich J, Nisenbaum R. Effect of Portable Rent Subsidies and Mentorship on Socioeconomic Inclusion for Young People Exiting Homelessness: A Community-Based Pilot Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2238670. doi: 10.1001/jamanetworkopen.2022.38670. PMID 36301546
- [Result] Thulien NS, Hwang SW, Kozloff N, Nisenbaum R, Akdikmen A, Fambegbe OP, Feraday R, Mathewson C, Mutamiri M, Roglich J, Wang A, Zagala M, Amiri A. "When I think about my future, I just see darkness": How youth exiting homelessness navigate the hazy, liminal space between socioeconomic exclusion and inclusion. Can J Public Health. 2023 Dec;114(6):893-905. doi: 10.17269/s41997-023-00804-2. Epub 2023 Jul 18. PMID 37462842
- [Derived] Thulien NS, Kozloff N, McCay E, Nisenbaum R, Wang A, Hwang SW. Evaluating the Effects of a Rent Subsidy and Mentoring Intervention for Youth Transitioning Out of Homelessness: Protocol for a Mixed Methods, Community-Based Pilot Randomized Controlled Trial. JMIR Res Protoc. 2019 Dec 20;8(12):e15557. doi: 10.2196/15557. PMID 31859688

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Started | 13 | 11
Completed | 11 | 11
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.5 (2.3) | 22.2 (2.1) | 21.8 (2.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 8 | 4 | 12
  Man | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black | 5 | 3 | 8
  Indigenous | 0 | 2 | 2
  White | 6 | 4 | 10
  Different choice | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 13 | 11 | 24
First time became homeless, age [Mean (Standard Deviation); unit: Years] | 18 (3.1) | 17.5 (4.3) | 17.8 (3.6)
Born in Canada [Count of Participants; unit: Participants] | 11 | 9 | 20
Immigration Status [Count of Participants; unit: Participants]
  Canadian citizen | 11 | 10 | 21
  Permanent resident | 1 | 1 | 2
  Refugee | 1 | 0 | 1
Child welfare involvement [Count of Participants; unit: Participants] — Participants were asked in the baseline survey whether the Children's Aid Society had ever been involved with them or their family. Participants who answered 'yes' have been reported here.
  Participants | 5 | 8 | 13
No. of attempts to live on own after being homeless [Count of Participants; unit: Participants] — Participants were asked in the baseline survey how many times they have tried to live on their own or with others after being homeless. Participant answers were grouped into 1-2 attempts or 3 or more attempts.
  Participants
    1-2 | 7 | 6 | 13
    ≥3 | 6 | 5 | 11
No. of attempts to exit homelessness [Count of Participants; unit: Participants] — Participants were asked in the baseline survey how many times they have attempted to exit homelessness. Participant answers were grouped into 1-2 attempts, 3-4 attempts, or 5 or more attempts.
  Participants
    1-2 | 7 | 6 | 13
    3-4 | 3 | 1 | 4
    ≥5 | 3 | 4 | 7
Highest educational level [Count of Participants; unit: Participants]
  Less than high school | 4 | 4 | 8
  Completed high school | 5 | 3 | 8
  Some or completed postsecondary education | 4 | 4 | 8
Regular contact with adult relative [Count of Participants; unit: Participants] — Participants were asked in the baseline survey if they are in regular contact with an adult relative (e.g., parent, grandparent, or aunt). Participants who answered 'yes' have been reported here.
  Participants | 12 | 7 | 19
Informal adult mentor [Count of Participants; unit: Participants] — Participants were asked in the baseline survey if they have an adult in their life whom they consider a mentor, and this mentor is not a relative and is outside of the social service sector. Participants who answered 'yes' have been reported here.
  Participants | 5 | 4 | 9
Employed [Count of Participants; unit: Participants] | 7 | 8 | 15
Social assistance [Count of Participants; unit: Participants] — Participants were asked in the baseline survey if they are receiving social assistance through Ontario Works or through the Ontario Disability Support Program.
  Participants
    Ontario Works | 8 | 4 | 12
    Ontario Disability Support Program | 2 | 4 | 6
ACEs, adverse childhood experiences [Count of Participants; unit: Participants] — Participants completed an adverse childhood experiences (ACEs) self-report questionnaire. A score of 4 or more is considered being at high risk for toxic stress. A score of 0 to 3 is considered being at a lower risk for toxic stress.
  Participants
    1-3 | 4 | 2 | 6
    4-9 | 8 | 9 | 17
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Community Integration Scale Score at 18 Months
Description: This outcome is a measure of behavioural (e.g., participation in activities) and psychological (e.g., sense of belonging) aspects of community integration. This will be measured using the Community Integration Scale (CIS), an 11-item scale. The CIS includes a psychological subscale (possible score range is from 4-20, 4 being low psychological community integration and 20 being high integration), and a physical subscale (total score range is 0-7, 0 being low physical community integration, and 7 being high integration). Only the psychological subscale has been reported here.
Time Frame: Change from baseline to 18 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 11.3 (2.6) | 10.8 (4.1)
  18 months | 11.2 (3.9) | 13.2 (2.9)
Statistical Analysis 1: Comparison: Rent Subsidies + Mentorship vs Rent Subsidies Only; Test type: Other; p = 0.18, ANCOVA; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-5.0 to 1.0]

2. Primary Outcome: Rosenberg Self-Esteem Scale Score at 18 Months
Description: This outcome is a measure of global self-worth and will be measured using the Rosenberg Self-Esteem Scale, a 10-item scale, internal consistency α = .77 - .88. The total scoring range is 0-30, a score of <15 is categorized as low self-esteem, and 15-30 is categorized as normal self-esteem.
Time Frame: Change from baseline to 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 16.0 (4.6) | 16.3 (6.1)
  18 months | 18.1 (5.2) | 19.6 (5.7)
Statistical Analysis 1: Comparison: Rent Subsidies + Mentorship vs Rent Subsidies Only; Test type: Other; p = 0.44, ANCOVA; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.0 to 2.3]

3. Secondary Outcome: Social Connectedness Scale Score at 18 Months
Description: This outcome is a measure of belongingness - the degree to which people feel connected to others. It is measured using the Social Connected Scale, a 20-item scale, internal consistency α = .92. The total scoring range is 20-120, 20 being low social connectedness and 120 being high social connectedness.
Time Frame: Change from baseline to 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 67.0 (12.9) | 77.0 (15.9)
  18 months | 74.2 (21.3) | 77.0 (25.8)
Statistical Analysis 1: Comparison: Rent Subsidies + Mentorship vs Rent Subsidies Only; Test type: Other; p = .38, ANCOVA; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [-9.7 to 24.4]

4. Secondary Outcome: Beck Hopelessness Scale Score at 18 Months
Description: This outcome is a measure of motivation, expectations, and feelings about the future and will be measured using Beck's Hopelessness Scale, a 20-item scale, internal consistency α = .93. The total scoring range is 0-20, 0-3 = None or minimal, 4-8 = Mild, 9-14 = Moderate - requires monitoring, 15+ = Severe - suicide risk.
Time Frame: Change from baseline to 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 4.5 (4.2) | 7.3 (4.8)
  18 months | 4.6 (4.8) | 5.8 (5.5)
Statistical Analysis 1: Comparison: Rent Subsidies + Mentorship vs Rent Subsidies Only; Test type: Other; p = 0.76, ANCOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-3.3 to 4.4]

5. Secondary Outcome: Academic/Vocational Participation as Assessed by a Questionnaire at 18 Months
Description: Participant engagement with school or a training program will be assessed. Participants will be prompted to answer questions about their current educational pursuit every 6 months in a questionnaire, including whether the individual is pursuing education, and the type of education.
Time Frame: Change from baseline to 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
Participants | 8 | 8
Statistical Analysis 1: Comparison: Rent Subsidies + Mentorship vs Rent Subsidies Only; Test type: Other; p = 0.68, ANCOVA

6. Other Pre Specified Outcome: Modified Engulfment Scale Score at 18 Months
Description: This is an exploratory outcome. This outcome is a measure of the degree to which an individual's self-concept is defined by their experience of homelessness. It will be assessed using the Modified Engulfment Scale, a 30-item scale, internal consistency α = .91. The total scoring range is 30-150, 30 being low engulfment, 150 being high engulfment. The scale was adapted for use in this study, substituting "experience of homelessness" for "illness". Increased levels of engulfment indicate that the individual was more likely to have an earlier age of onset (of homelessness), to have experienced a longer period of homelessness, with a greater number of homelessness/shelter contact, and a decreased level of social adjustment.
Time Frame: Change from baseline to 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 81.6 (13.6) | 83.8 (28.1)
  18 months | 70.4 (15.3) | 79.5 (27.0)
Statistical Analysis 1: Comparison: Rent Subsidies + Mentorship vs Rent Subsidies Only; Test type: Other; p = 0.12, ANCOVA; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-16.4 to 2.0]

7. Other Pre Specified Outcome: Modified Colorado Symptom Index Score at 18 Months
Description: This is an exploratory outcome; it is the measurement of the presence and frequency of psychiatric symptoms experienced in the past month. Measured using the Modified Colorado Symptom Index, a 14-item questionnaire, internal consistency α = .90 - .92. The total scoring range is 0-56, 0 being a low frequency of psychiatric symptoms, and 56 being a high frequency of psychiatric symptoms.
Time Frame: Change from baseline to 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 40.9 (10.6) | 36.8 (15.4)
  18 months | 32.9 (10.0) | 34.9 (16.0)
Statistical Analysis 1: Comparison: Rent Subsidies + Mentorship vs Rent Subsidies Only; Test type: Other; p = 0.34, ANCOVA; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-13.7 to 5.0]

8. Other Pre Specified Outcome: Income as Assessed by a Questionnaire at 18 Months
Description: This is an exploratory outcome. Participants will be prompted to answer questions about their current income every 6 months in a questionnaire. This outcome is assessed using a repeated measures analysis and changes in income will be assessed for change over time at the aggregate level.
Time Frame: Change from baseline to 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
Participants
  Receiving Employment Income at Baseline | 7 | 8
  Receiving Employment Income at 18 Months | 5 | 5

9. Other Pre Specified Outcome: Perceived Housing Quality Scale Score at 18 Months
Description: This is an exploratory outcome and is assessed by participant perception of housing choice and quality. Measured using the Perceived Housing Quality Scale.This scale was used extensively in the Chez Soi/At Home study, but psychometric properties have yet to be reported. It has been shortened it from 10 items (Chez Soi/At Home) to seven relevant items. The total scoring range is 7-35, 7 being very dissatisfied with current housing quality, and 35 being very satisfied with housing quality.
Time Frame: Change from baseline to 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 24.6 (4.1) | 23.5 (5.2)
  18 months | 23.8 (6.1) | 24.6 (6.6)
Statistical Analysis 1: Comparison: Rent Subsidies + Mentorship vs Rent Subsidies Only; Test type: Other; p = 0.62, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-6.6 to 4.0]

10. Other Pre Specified Outcome: Barriers and Facilitators of Social and Economic Inclusion: Key Themes and Subthemes as Informed by Individual Interviews With Youth Participants at 30 Months
Description: This is an exploratory outcome. Using one-on-one, semi-structured interviews with young people from both the control and intervention arms, we examined and compared their experiences of social and economic inclusion. Additionally, we explored how mentorship, provided to youth in the intervention arm, influenced this experience.
Time Frame: Assessed every 6 months for 30 months, starting at baseline.
Population: Participants from both groups were included to explore factors beyond the intervention impacting socioeconomic inclusion. The path to inclusion is complex, with factors like informal mentorship (from non-study mentors) proving more influential than formal study mentorship. Thus, analyzing the groups as a cohort provided a more comprehensive understanding of participants' experiences.
Measure: Number; unit: Key themes and sub-themes
Groups:
- Pooled Analysis of Intervention and Control Groups: Data for the intervention and control groups were pooled.
Arm/Group | Pooled Analysis of Intervention and Control Groups
Number analyzed (Participants) | 12
Key themes and sub-themes
  Themes | 3
  Subthemes | 10

11. Other Pre Specified Outcome: Barriers and Facilitators of Mentorship Intervention: Key Themes and Subthemes as Informed by Focus Groups With Mentors at 24 Months
Description: This is an exploratory outcome. We conducted focus groups with study mentors to explore their perception of barriers and facilitators to mentorship engagement.
Time Frame: Assessed at 12 and 24 months.
Population: Mentors that were matched with youth in the intervention arm.
Measure: Number; unit: Key themes and sub-themes
Groups:
- Mentors: Data from study mentors.
Arm/Group | Mentors
Number analyzed (Participants) | 9
Key themes and sub-themes
  Themes | 3
  Sub-themes | 11

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Rent Subsidies + Mentorship | Rent Subsidies Only
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03779204/Prot_SAP_000.pdf